CLINICAL TRIAL: NCT03658616
Title: Combined Randomized, Double-blind, Dose-confirming Phase 3a Study in Parallel Design to Assess the Efficacy and Safety of Topical 4-week Treatment With 1% GPB Cream vs Placebo and Open-label Phase 3b Study to Assess Long-term Efficacy and Safety in Patients With Primary Axillary Hyperhidrosis Treated With 1% GPB Cream
Brief Title: Assessment of Efficacy and Safety of Topical Administration of 1% Glycopyrronium Bromide (GPB) in Patients With Primary Axillary Hyperhidrosis and the Assessment of Long-term Efficacy and Safety of Topical Administration of 1% GPB Cream in Patients With Primary Axillary Hyperhidrosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hyp1-18/2016
Record Dates: First submitted 2018-09-03; First posted 2018-09-05 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Excessive sweating
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WO3970 (Experimental): Formulation containing WO3979 for topical application
  Interventions: Drug: WO3970
- Placebo of WO3988 (Placebo Comparator): Formulation containing Placebo of WO3988 for topical application
  Interventions: Drug: Placebo (WO3988)

INTERVENTIONS:
Drug: WO3970 — Application of cream to each axilla
  Arms: WO3970
Drug: Placebo (WO3988) — Application of cream to each axilla
  Arms: Placebo of WO3988

SUMMARY:
The aim of this study is to investigate the efficacy and safety of 1% GPB cream after 4 weeks of treatment compared with placebo with a sufficient number of patients to obtain statistically significant results, and to assess the long-term safety of 1% GPB cream.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe primary axillary hyperhidrosis with a HDSS score of 3 or 4
* At least 50 mg of sweat production in each axilla measured gravimetrically at room temperature and at a humidity consistent with the normal climate in that area over a period of 5 minutes (patients should have acclimatized to that room for at least 30 minutes)
* Men and women aged 18 to 65 years at the time of informed consent with a body mass index of 18-32 kg/m2
* Able to comply with protocol requirements, including overnight stays, blood sample collections as defined in the protocol subjects
* Willing and able to provide written informed consent

Exclusion Criteria:

* Known allergy to any of the components in the investigational product.
* Hypersensitivity against glycopyrrolate
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria, climacteric hyperhidrosis.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Botulinum toxin treatment in the prior 4 months.
* Angle closure glaucoma or its precipitation (narrow angle).
* Mycotic, other skin infections and other dermal disorder including infection at anticipated application sites in either axilla.
* Any condition or situation that, in the investigator's or sub-investigator's opinion, may interfere with the patient's participation in the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Dose-confirming part: Absolute change in sweat production assessed by gravimetric measurement (GM) from Baseline (Day 1a) to Day 29 in the 1% GPB group compared with the placebo group. | Baseline (Day 1a), Day 29
Long-term part (only for newly recruited patients): Absolute change in sweat production assessed by GM from Baseline (Day 1b) to Week 12 | Baseline (Day 1b), Week 12

SECONDARY OUTCOMES:
Dose-confirming part: Percentage of responders assessed by the Hyperhidrosis Disease Severity Scale (HDSS) (≥2-point improvement from Baseline) on Day 29 in the 1% GPB group compared with the placebo group | Day 29
  The Hyperhidrosis Disease Severity Scale (HDSS) is a disease-specific, quick, and easily-understood diagnostic tool that provides a qualitative measure of the severity of the patient's condition based on how it affects daily activities. HDSS is a four item scale. A score of 1 or 2 indicates mild or moderate Hyperhidrosis. A score of 3 or 4 indicates severe Hyperhidrosis.
Dose-confirming part: Percentage of responders assessed by GM at Day 29 (defined by sweat reduction of ≥50%, ≥75%, and ≥90% compared with Baseline) in the 1% GPB group compared with the placebo group | Day 29
Long-term part: Percentage of responders assessed by the HDSS (≥2-point improvement from Baseline) at Week 12 | Week 12
Long-term part: Percentage of responders assessed by GM at Week 4 and Week 12 (defined by sweat reduction of ≥50%, ≥75%, and ≥90% compared with Baseline | Week 4, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rolf-Markus Szeimies, MD, Principal Investigator — Klinikum Vest GmbH, Knappschaftskrankenhaus Recklinghausen
Locations (1):
- Dr. Harald Brüning, Kiel, Germany

REFERENCES:
- [Derived] Donhauser T, Apfelbacher C, Kann G, Masur C, Kamudoni P, Salek S, Abels C, Gabes M. Hyperhidrosis quality of life index (HidroQoL): further validation by applying classical test theory and item response theory using data from a phase III clinical trial. J Patient Rep Outcomes. 2023 Jun 6;7(1):55. doi: 10.1186/s41687-023-00596-6. PMID 37280417